CLINICAL TRIAL: NCT00306943
Title: Phase III Vaccination Study for Evaluation of Immunogenicity and Reactogenicity of Influsplit SSW 2004/2005 in People Age 18 or Beyond
Brief Title: Annual Study for Fluarix Registration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104745
Record Dates: First submitted 2005-09-15; First posted 2006-03-27 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Influsplit SSW®

SUMMARY:
A pre-requisite to the yearly licensing process of the Influenza vaccine (FluarixTM/ Influsplit SSW®) is to demonstrate in clinical studies, the immunogenicity and reactogenicity of the vaccine composed of the new strains (2005/2006).

DETAILED DESCRIPTION:
Since 1998 it is common practice within the European Community, to grant new licensees for Influenza Vaccines including the actual strain composition, by realizing the EU "Mutual Recognition Procedure" The procedure foresees the clinical testing of the vaccine before approval according to the particulars in the EU-Document CPMP/BWP/214/96: "Note for Guidance on Harmonization of Requirements for Influenza Vaccines" of the "Committee for Proprietary Medical Products (CPMP) as Sub-Organization of the "European Agency for the Evaluation of Medicinal Products". Assessment of the Immunogenicity and Reactogenicity of the in its strain composition actualized, Influenza split vaccine2004/2005 (Influenza split vaccine 2005/2006) versus the criteria of the CPMP.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return, and follow-up visits) should be enrolled in the study.
* All Subjects, enrolled in this study, must not been immunized against Influenza within the season 2003/2004.
* Written informed consent obtained from the subject must be available, after the subject has been informed in an understandable language.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e., oral temperature / axillary temperature <37.5°C (99.5°F).
* Acute clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Pregnancy (exclusion by safe contraception; pregnancy test at day 0.
* Known allergic reactions, probably caused by one or more vaccine ingredients.
* Drug and/or Alcohol abusers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Investigation of the humoral immune response (haemagglutination inhibiting antibodies) in subjects

SECONDARY OUTCOMES:
Investigation of the safety and reactogenicity in subject's age 18 or elder past application of a doses of Influenza split vaccine 2005/2006 in relation to solicited and non-solicited incidents.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register